CLINICAL TRIAL: NCT00552721
Title: Physical Therapy With Versus Without Strength Training After Botulinum-toxin Treatment in Children With Cerebral Palsy
Brief Title: Physical Therapy After Anti-spastic Treatment in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KF 02 323948
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Last update posted 2009-09-07 (Estimated); Status verified 2009-09

CONDITIONS: Cerebral Palsy
Keywords: Motor control; Spasticity
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — Physical Therapy Modalities; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Physical therapy with strength training.
  Interventions: Other: Physical therapy with strength training
- B (Active Comparator): Physical therapy without strength training.
  Interventions: Other: Physical therapy without strength training

INTERVENTIONS:
Other: Physical therapy with strength training — 12 weeks of physical therapy after Botulinum-toxin treatment (two 45-min sessions/week) with an emphasis on strength training.
  Arms: A
Other: Physical therapy without strength training — 12 weeks of physical therapy after Botulinum-toxin treatment (two 45-min sessions/week) without strength training.
  Arms: B

SUMMARY:
It is the primary purpose of this pilot study to investigate if physical therapy with strength training is better at improving muscle and gait function after anti-spastic treatment with Botulinum toxin compared to physical therapy without strength training in children with cerebral palsy. The investigators hypothesize that it is.

ELIGIBILITY:
Inclusion Criteria:

* cerebral palsy (diplegia and hemiplegia)
* indication for anti-spastic treatment with Botulinum toxin

Exclusion Criteria:

* fixed contractures

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2007-10; Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Three-dimensional gait analysis | 12 weeks
Selective motor control | 12 weeks

SECONDARY OUTCOMES:
Spasticity (modified Ashworth) | 12 weeks
Range of motion | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bandholm, MSc, Principal Investigator — Gait Analysis Laboratory, Department of Orthopedic Surgery, Hvidovre University Hospital; Stig Sonne-Holm, MD, DSc, Study Chair — Gait Analysis Laboratory, Department of Orthopedic Surgery, Hvidovre University Hospital; Bente R Jensen, PhD, Study Chair — Institute of Exercise and Sport Sciences, University of Copenhagen; Søren A Pedersen, MD, Study Chair — Hvidovre University Hospital
Locations (1):
- Gait Analysis Laboratory, Department of Orthopedic Surgery, Hvidovre University Hospital, Hvidovre, Denmark